CLINICAL TRIAL: NCT00722839
Title: A Phase I Dose Escalation Study of Peptide Vaccines With Activity Against Human Cytomegalovirus
Brief Title: Vaccine Therapy in Preventing Cytomegalovirus in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: City of Hope Medical Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: City of Hope 03121; R01CA077544 (NIH); P30CA033572 (NIH); CHNMC-03121; CDR0000599724 (Registry Identifier: NCI PDQ); NCI-2010-01227 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2008-07-25; First posted 2008-07-28 (Estimated); Last update posted 2012-06-25 (Estimated); Status verified 2012-06

CONDITIONS: Nonneoplastic Condition
Keywords: cytomegalovirus infection
MeSH Terms: conditions — Cytomegalovirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group A (Experimental): Participants receive either PADRE-CMV fusion peptide vaccine or tetanus-CMV fusion peptide vaccine subcutaneously (SC) on days 1, 21, 42, and 63 in the absence of unacceptable toxicity.
  Interventions: Biological: PADRE-CMV fusion peptide vaccine; Biological: tetanus-CMV fusion peptide vaccine
- Group B (Experimental): Participants receive either PADRE-CMV fusion peptide vaccine in CpG 7909 adjuvant SC or tetanus-CMV fusion peptide vaccine in CpG 7909 adjuvant SC on days 1, 21, 42, and 63 in the absence of unacceptable toxicity.
  Interventions: Biological: PADRE-CMV fusion peptide vaccine; Biological: tetanus-CMV fusion peptide vaccine; Drug: agatolimod sodium

INTERVENTIONS:
Biological: PADRE-CMV fusion peptide vaccine — Given subcutaneously
Biological: tetanus-CMV fusion peptide vaccine — Given subcutaneously
Drug: agatolimod sodium — Given subcutaneously
  Arms: Group B

SUMMARY:
RATIONALE: Vaccines made from peptides may help the body build an immune response to kill cytomegalovirus.

PURPOSE: This phase I trial is studying the side effects and best dose of vaccine therapy in preventing cytomegalovirus in healthy participants.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* To establish whether 3 vaccine dose levels of PADRE-CMV and tetanus-CMV fusion peptide vaccines are safe and well tolerated in healthy cytomegalovirus (CMV)-seropositive or -seronegative participants.
* To establish safe dose levels for the PADRE-CMV and tetanus-CMV fusion peptide vaccines in combination with PF 03512676 DNA in these participants.

Secondary

* To provide preliminary evidence of enhanced cellular immunity to CMV at levels of T cells that would support potential feasibility if such cells were to be transferred from the donor to recipients of hematopoietic stem cell transplantation (HSCT) in amounts consistent with protection against disease.
* To determine whether a reduced dose of peptide vaccine can be immunogenic in combination with PF 03512676 DNA.
* To confer CMV-specific cytotoxic T-lymphocyte (CTL) function to CMV-negative participants.
* To determine the duration of immune enhancement of CMV-specific CTL function up to 12 months following immunization of healthy participants.

OUTLINE: This is a dose-escalation study of PADRE-CMV and tetanus-CMV fusion peptide vaccines. Participants are stratified according to cytomegalovirus (CMV) serum status (positive vs negative). Participants are assigned to 1 of 2 groups.

* Group A: Participants receive either PADRE-CMV fusion peptide vaccine or tetanus-CMV fusion peptide vaccine subcutaneously (SC) on days 1, 21, 42, and 63 in the absence of unacceptable toxicity.
* Group B: Participants receive either PADRE-CMV fusion peptide vaccine in CpG 7909 adjuvant SC or tetanus-CMV fusion peptide vaccine in CpG 7909 adjuvant SC on days 1, 21, 42, and 63 in the absence of unacceptable toxicity.

Participants are contacted by telephone every 3-7 days after immunization. Participants also complete a notebook on any health-related event for 14 days after each immunization.

Participants undergo blood sample collection at baseline and periodically during study for immunologic laboratory studies, including flow cytometry, by HLA-A2-CMV-tetramer, CMV-specific intracellular cytokine, CMV-specific CD107 degranulation, lymphoproliferation, and chromium release assays.

After completion of study therapy, participants are followed for up to 1 year.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Cytomegalovirus (CMV) seropositivity or seronegativity
* HLA A*0201 positive OR positive tetramer-binding using CMV peptide 495-503 with HLA A2 subtypes other than HLA A*0201
* A2-CMV-Tet cells ≤ 10^8/L

PATIENT CHARACTERISTICS:

* Platelet count within 1.5 times upper level of normal (ULN)
* The following blood and chemistry studies must be normal:

  * Sodium
  * Potassium
  * Chloride
  * Carbon dioxide
  * Glucose
  * BUN
  * Creatinine
  * Uric acid
  * WBC
  * Hemoglobin
  * Hematocrit
* The following studies must be ≤ ULN:

  * Albumin
  * Alkaline phosphatase
  * AST and ALT
  * Lactic dehydrogenase
  * Total bilirubin
* Hepatitis B virus surface antigen negative
* Hepatitis C virus seronegative
* No diagnosis that is associated with immunodeficiency (e.g., HIV)
* No active infection that requires treatment
* No known cardiac disease including hypertension and/or high cholesterol
* No serious abnormalities by EKG (in participants ≥ 50 years of age)
* Not pregnant
* Negative pregnancy test
* Fertile participants must use effective contraception during study and for 6 weeks after the fourth and last dose of vaccine
* No history of allergic reaction to tetanus toxoid
* No history of any of the following:

  * Cancer other than basal cell carcinoma of the skin
  * Depression
  * Allergic diathesis, as defined by a history of asthma
  * Anaphylaxis
  * Generalized urticaria or daily use of antihistamines
  * Episodic (more than once in the past 3 months) inhalational medications including steroidal agents
  * Non-steroidal agents or cromolyn sodium
  * Frequent migraines, defined as 3 or more episodes in the past year
* No prior or concurrent infectious condition

PRIOR CONCURRENT THERAPY:

* More than 6 months since prior participation in a CMV immunotherapy trial
* More than 30 days since prior live vaccine
* More than 2 weeks since prior inactivated vaccine
* No concurrent daily medications for chronic or current illness, except for the following:

  * Thyroid-replacement therapy
  * Estrogen-replacement therapy
  * Dietary vitamins and protein supplements
  * Any medication, as determined by the principal investigator, that is not known or likely to be immunosuppressive
* No surgery in the past 6 months that required general anesthesia

  * Minor procedures (e.g., dental surgery or superficial diagnostics biopsies) allowed

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 68 (Actual)
Dates: Start 2006-12; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Successful completion of a series of 4 injections (at weeks 0, 3, 6, and 9) without dose-limiting toxicity | 3 weeks after the final vaccine dose
Maximum tolerated dose of each vaccine with or without adjuvant CpG 7909 | 1 year after the final vaccine dose

SECONDARY OUTCOMES:
Number of CMV-positive and CMV-specific CD8+ T cells/L | 1 year after final vaccine dose

CONTACTS AND LOCATIONS:
Overall Officials: John A. Zaia, MD, Principal Investigator — City of Hope Comprehensive Cancer Center
Locations (1):
- City of Hope Comprehensive Cancer Center, Duarte, California, United States

REFERENCES:
- [Derived] La Rosa C, Longmate J, Lacey SF, Kaltcheva T, Sharan R, Marsano D, Kwon P, Drake J, Williams B, Denison S, Broyer S, Couture L, Nakamura R, Dadwal S, Kelsey MI, Krieg AM, Diamond DJ, Zaia JA. Clinical evaluation of safety and immunogenicity of PADRE-cytomegalovirus (CMV) and tetanus-CMV fusion peptide vaccines with or without PF03512676 adjuvant. J Infect Dis. 2012 Apr 15;205(8):1294-304. doi: 10.1093/infdis/jis107. Epub 2012 Mar 7. PMID 22402037